CLINICAL TRIAL: NCT07148297
Title: Proof-of-concept Case-control Study for Colorectal Cancer Assessment Using Delta-HLD Technology (CASCADE)
Brief Title: Colorectal Analysis for Signature Cancer Assessment Using Delta-HLD
Acronym: CASCADE
Status: Recruiting | Type: Observational
Sponsor: Epiliquid Holding, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CRC-CPOC; RENIS IS003779 (Other: Epiliquid Holding, Inc)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-08

CONDITIONS: Colo-rectal Cancer
Keywords: Colorectal cancer; Epigenetics; Liquid Biopsy; cfDNA; Biomarker; Methylation; PCR
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma (cfDNA) samples collected from whole blood, tumor tissue samples (formalin-fixed or fresh-frozen) and normal colonic tissue collected from colorectal cancer patients at the time of diagnosis. Plasma samples will also be retained from colonoscopy-negative controls. All specimens will be used for biomarker analysis using delta-HLD technology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRC Cases: Individuals with histologically confirmed colorectal adenocarcinoma
- Controls: Individuals with negative colonoscopy results and no history of colorectal cancer

SUMMARY:
CASCADE (Colorectal Analysis for Signature Cancer Assessment Using delta-HLD Technology) is a proof-of-concept case-control study designed to evaluate the performance of delta-HLD, Epiliquid's proprietary liquid biopsy technology, for the detection of colorectal cancer. Epiliquid also integrates a proprietary bioinformatic system capable of identifying, ranking, and selecting tumor-specific methylation biomarkers for different cancer types. In this study, colorectal cancer-specific biomarkers will be evaluated in blood and tissue samples using delta-HLD technology, which enables sensitive and multiplexed detection through PCR. Study results will support the validation of Epiliquid's integrated platform as a minimally invasive and accessible diagnostic solution for colorectal cancer.

DETAILED DESCRIPTION:
This observational case-control study aims to evaluate the performance of delta-HLD technology in an average-risk colorectal cancer population. The CASCADE study seeks to validate the technical and diagnostic performance of Epiliquid's platform, which integrates a proprietary bioinformatic system designed to identify, rank, and select methylation-based biomarkers specific to each cancer type. For colorectal cancer, these biomarkers are selected and detected using delta-HLD technology, a proprietary method that combines sequential enzymatic pre-treatment with PCR-based amplification to enable sensitive, multiplexed detection. Blood (plasma cfDNA) and tumor tissue samples will be collected from two groups: individuals with histologically confirmed colorectal cancer (cases) and individuals with negative colonoscopy findings (controls). This proof-of-concept study will assess biomarker performance, including sensitivity, specificity, and concordance between blood and tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for colonoscopy or colorectal surgery
* Willing and able to provide informed consent
* Able to provide blood and/or tissue sample before treatment or resection

Exclusion Criteria:

* Prior history of colorectal cancer
* Inflammatory bowel disease
* Known hereditary cancer syndromes (e.g., Lynch, FAP)
* Other active malignancies
* Recent chemotherapy or immunosuppressive treatment

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 45 to 75 years from an average-risk population for colorectal cancer, undergoing colonoscopy or colorectal surgery at participating clinical sites in Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of delta-HLD Technology for Colorectal Cancer | Within 3 months after sample collection
  Diagnostic performance of methylation biomarkers detected using delta-HLD technology in plasma and tissue samples, using colonoscopy and histopathology as the clinical reference standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Epiliquid, Mendoza, Argentina

IPD SHARING:
Plan to Share IPD: No